CLINICAL TRIAL: NCT06207227
Title: A Feasibility Study to Evaluate the Clinical Performance and Safety of the VITA AV Clinical System When Used for the Treatment of Vaginal Atrophy
Brief Title: Clinical Performance and Safety of the VITA AV Clinical System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AVeta Medical (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10545
Record Dates: First submitted 2023-12-13; First posted 2024-01-16 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Vaginal Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VITA AV Clinical System (Experimental): VITA AV Clinical System
  Interventions: Device: VITA AV Clinical System

INTERVENTIONS:
Device: VITA AV Clinical System — The VITA AV Clinical System that works on the principle of negative pressure suction to the vaginal wall to treat VA, based on the idea of the clinical application in wound healing which is intended to elicit improvements in the rate of angiogenesis, moisture and HA production post-treatment. It is believed that the VITA AV Clinical System will provide a more effective treatment by improving the underlying cellular deficiencies associated with VA.

SUMMARY:
The primary objective of this clinical investigation is to demonstrate that treatment with the VITA AV clinical system is feasible and to evaluate clinical performance and safety when used to improve the symptoms and signs of vaginal atrophy (VA) due to menopause.

DETAILED DESCRIPTION:
After recruitment of the subject, the initial assessment of the enrolled patient will be performed, which includes screening, baseline evaluations & pre-procedural assessments, suitability of device size for each patient (vaginal dilator kit- for sizing and recording) and endoscopic images will be done by the clinician.

Subjects will be introduced to the therapy over a 2-4week familiarisation period to determine their dosage. Subsequently, subjects will receive 3x treatment sessions over a 12-week window with a final follow-up 4 weeks after the final treatment session.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy postmenopausal women from 51 years up to and including 70 years.
2. The subject must be able to identify an MBS of at least moderate severity from one of the following: vaginal dryness, itching, discharge, and dyspareunia (pain during intercourse).
3. Vaginal Health Index (VHI) score between 6-15, indicating mild to moderate VA.
4. The one-size intravaginal tip "VITA AV probe Kit" fits comfortably within the subject's vagina. Clinician to size the vagina using the vaginal dilator sizing kit and record the size on the assessment/record sheet. (25mm diameter, 60mm length). Urethral opening is distal to device sealing collar.
5. Normal Papanicolaou test within the past year (or should be done before the trial begins or 2 weeks before F1). Subject can ONLY participate on negative results.
6. Vaginal canal free of any lesions or abnormalities other than signs of VA.
7. Willing and able to sign an Informed Consent Form (ICF).
8. Subjects must be willing to refrain from sexual intercourse for 48 hours before initial assessment, for 48 hours before and after each session [Familiarisation (F) and Treatment (T)] and for 48 hours before final follow-up visit.
9. Subjects must be willing to stop using any lubricant at least 48hrs before initial assessment (as if they use lubricant, it will affect sizing)before and after each session [Familiarisation (F) and Treatment (T)] and for 48 hours before final follow-up visit. Only use lubricant provided by the clinic to aid sexual intercourse
10. Subjects must be willing to discontinue/stop dilator/pelvic floor therapy 7 days before initial assessment and this therapy should not continue if the patient is participating in trial.

Exclusion Criteria:

1. Vaginal Health Index (VHI) score of 5 or less (indicates severe VA).
2. Subjects on Hormone Replacement Therapies (HRT), systemic or local, or within 6 months of cessation of HRT prior to inclusion in the study.
3. Use of vaginal moisturisers, or any other local vaginal preparation within 3 months prior to study inclusion.

   Note: The use of simple non-moisturising lubricants to aid sexual intercourse can be accepted in the study.
4. Subjects with bleeding disorders.
5. Subjects on prescribed blood thinners such as antiplatelets and anticoagulants (Heparins, Warfarin or Clopidogrel).
6. Acute UTIs.
7. Any active genital infections.
8. Abnormal Pap smear test.
9. Positive pregnancy test or planned pregnancy during the study period.
10. Uterine prolapse.
11. Subjects with urogenital sinus (this is when urethral opening is combined with the vagina opening), otherwise the urethral opening will be traumatized resulting in an UTI.
12. Undergone pelvic surgery within 6 months prior to the start of the study.
13. Undiagnosed vaginal bleeding.
14. Cancer patients on chemotherapy or subjects with any diagnosed gynaecological cancers.
15. Breast cancer survivors who have had chemotherapy within the last 5 years or are on aromatase inhibitors.
16. Subjects where the one-size VITA AV intravaginal tip does not fit comfortably within the patient's vagina (in the clinician's opinion).
17. Any serious disease or chronic condition that could jeopardize the subject's ability to complete the trial assessments.
18. Subjects who, in the opinion of the investigator, will be inappropriate for inclusion in this study or will not comply with the requirements of the study.
19. Subjects who do not have the mental or physical ability to comply with time schedules and further study procedures.
20. Subjects with urinary symptoms as their MBS will be excluded from the study due to other potential causes of this symptom.

Ages: 51 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-04-13 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Most Bothersome Symptom (MBS) Improvement from Baseline to 1-Month Follow-Up | Follow-Up Visit at 1 month
  To demonstrate that treatment with the VITA AV Clinical System improves the Most Bothersome Symptom (MBS) of VA in more than 50% of subjects after 3 treatment sessions at MTD.
  The MBS is selected from a list of symptoms (including vaginal dryness, itching, discharge, and dyspareunia (pain during intercourse)) and the subject must select a single symptom (among those classified as moderate to severe) as the MBS.
  MBS assessment (using a severity rating of no symptom, mild, moderate, severe) will be completed at baseline and immediately before each treatment session and 4 weeks after the last session during the follow-up phase. The change in the severity of the MBS from baseline to the 4-weeks after the last treatment is the evaluation for symptomatic improvement.
Primary Safety Endpoint #1:The degree of pain experienced during each treatment session from the first to the last treatment. | Lat Treatment
  The degree of pain experienced during each treatment session will be assessed by using visual analogue scale (VAS), where the left extreme indicates 'no pain or discomfort', and the right extreme indicates 'severe pain or discomfort'.
Primary Safety Endpoint #2: Serious Adverse Events (SAEs) | Follow-Up Visit at 1 month
  Assessment of Serious Adverse Events (SAEs) with emphasis on device or treatment related events.
Primary Safety Endpoint #3: Serious Adverse Device Effects (SADEs) at each treatment and follow-up visit. | Follow-Up Visit at 1 month
  Serious Adverse Device Effects (SADEs) with emphasis on device or treatment related events.

SECONDARY OUTCOMES:
Vaginal Maturation Index (VMI) Improvement | Final Follow-Up Visit at 1 month
  Percent improvement in Vaginal Maturation Index (VMI) from the initial assessment visit to the final follow-up visit/session is calculated at 4 weeks after the last treatment and at the final follow-up visit.
  VMI Score is assigned as follows:
  1. ☐ 65% - 100% (premenopausal women with estrogenic environment).
  2. ☐ 50% - 64% (Moderate zero estrogenic effects on cells).
  3. ☐ ≤ 49% (zero estrogenic effects on cells).
  An increase in VMI score is expected.
Vaginal/urinal pH Improvement | Final Follow-Up Visit at 1 month
  Improvement in vaginal/urinal pH from the initial assessment visit to after 3x treatment sessions at MTD and at the final follow-up visit.
Vaginal Health Index (VHI) Improvement | Follow-Up Visit at 1 month
  Percent improvement in the Vaginal Health Index score (VHI) from the initial assessment visit to after 3x treatment sessions at MTD and at the final follow-up visit.
  VHI score is assigned as follows:
  1. ☐ 6 - 8.
  2. ☐ 9 - 12.
  3. ☐ 13 - 15.
  4. ☐ MORE THAN 15.
  An increase in VHI score is expected.
Improvement in visual appearance of the vaginal mucosa | Follow-Up Visit at 1 month
  Improvement in visual appearance of the vaginal mucosa (as assessed by endoscopic images) from the initial assessment visit to 4 weeks after the last treatment has been delivered.
Overall subject satisfaction with treatment after 3x treatment sessions at MTD at the final follow-up visit | Follow-Up Visit at 1 month
  Overall subject satisfaction with treatment after 3x treatment sessions at MTD at the final follow-up visit. The subject answers the following question 'Taking into account changes in VA symptoms, in overall well-being and quality of life, and any adverse events experienced, how would you define your level of satisfaction with the treatment and the device?'
  Overall subject satisfaction is subjective based on the subject's experience and is assigned the following rating:
  1. ☐ POOR
  2. ☐ FAIR
  3. ☐ GOOD
  4. ☐ VERY GOOD
  5. ☐ EXCELLENT

OTHER OUTCOMES:
Long Term Safety Data (Trial Extension) | Follow-Up Visit at 12 month
  Evaluation of Adverse Events (serious and non-serious) at 12 months post final treatment
Long Term Clinical Effect (Trial Extension) | Follow-Up Visit at 12 month
  Evaluation of the long-term clinical effect based on subjective evidence for symptom relief experienced as a result of the VITA AV Clinical System treatment, i.e., the severity rating of the MBS as indicated by the subject at the 10- and 12-month follow-up visits.
Long Term Durability (Trial Extension) | Follow-Up Visit at 12 month
  Durability of benefit of the VITA AV treatment is assessed based on the subjects' answers to the following question "From the final treatment, approximately how long did the benefit/improvement last?" which is gathered at the 10- and 12-month follow-up visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Pineo Clinic (Pineo Medical Ecosystem), Tbilisi, Georgia

IPD SHARING:
Plan to Share IPD: No